CLINICAL TRIAL: NCT01023620
Title: Human Immunodeficiency Virus Acquired Lipodystrophy (HAL) Classification, Measurement, & Fat Response to a Thiazolidinedione (TZD) Challenge in Differing Adult Phenotypic Presentations
Brief Title: HIV Acquired Lipodystrophy (HAL) Classification, Measurement and Fat Response to Thiazolidinedione (TZD) (Pioglitazone)
Acronym: HAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Takeda IISR - MSA-PIO-028
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: HIV Infections
Keywords: HIV; Lipodystrophy; Lipoatrophy; Lipohypertrophy; Human Immunodeficiency Virus
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Acquired Immunodeficiency Syndrome | interventions — Pioglitazone; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Experimental): 10 male patients with lipodystrophy taking daily Pioglitazone 45 mg
  Interventions: Drug: Pioglitazone
- Observation/Comparison (Sham Comparator): 10 male patients with lipodystrophy not taking daily Pioglitazone
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Pioglitazone — Participants will take oral Pioglitazone 45 mg daily for 16 weeks.
  Other Names: Actos
  Arms: Pioglitazone
Other: Observation — Participants will be observed for 16 weeks but will not receive drug
  Other Names: Comparison
  Arms: Observation/Comparison

SUMMARY:
This study is being done to better understand why people with HIV who have taken drugs for HIV begin to show abnormal changes in fat loss or fat gain in their bodies. This condition is called lipodystrophy.

Patients who take medicine for HIV and who have lipodystrophy report loss of subcutaneous (sc) fat from the arms, legs, and face and excess fat gain in the neck and truncal region. They also more likely to have problems with insulin in the body, high fat levels in the blood and diabetes. The reason that lipodystrophy develops is not fully understood although some HIV drugs have are very likely the cause. The complications pose an increased risk of fat blockage forming in the arteries making you more at risk for heart problems in the future. Changes in body fat can cause physical discomfort and psychological distress. Management of these problems can be a challenge for the patient's doctor.

The investigators propose data collection to determine if there is more than one reason why this might happen in some people and not in others. Laboratory samples being collected: 1) special imaging of the liver; 2) fat collected by needle from the mid thigh and mid-shoulder areas; 3) blood samples to measure the virus, t-cells, fats, and other markers of how the patient's body is handling the virus.

This study is being done because science does not fully understand why some patients with HIV who take medicines for the virus have abnormal fat loss or gain and some do not. This research study is intended to help us better understand why and how this happens.

ELIGIBILITY:
Inclusion Criteria:

Participants must be 18 years of age or older of all racial and ethnic origins, and capable of giving informed consent. Spanish speaking individuals are eligible for participation.

Additionally they must be/have:

1. Biologically male (not transgendered)
2. HIV positive for at least 24 months,
3. On stable HAART for at least the last 3 months prior to entering the study,
4. Practitioner diagnosed lipodystrophy as defined by:

aHAL (any of these) decreased subcutaneous fat in the limbs with prominent veins, loss of buttock fat or facial atrophy hHAL: fat accumulation in abdomen and/or dorsocervical region

Exclusion Criteria:

Participants cannot be less than 18 years of age, institutionalized, nor have prior diseases or conditions that may alter body fat composition. Exclusions:

1. Females are excluded
2. Prior history of CHF
3. Prior history of macular retinal edema
4. Prior history of spontaneous bone fracture
5. Diabetics receiving oral/injected/inhaled diabetic agents or individuals with a fasting blood glucose value greater than or equal to 140 within the last 90 days.
6. Current active opportunistic infections for example :

   1. PCP pneumonia
   2. Neuropathy
   3. Thrush
   4. Systemic KS (Kaposi sarcoma)

   i) localized cutaneous lesions are not an exclusion e) MAC (Mycobacterium Avium complex) f) Histoplasmosis g) Coccidioidomycosis
7. Planning to discontinue HAART
8. Current diagnosis of cancer or receiving chemotherapy
9. Systemic steroid use during the prior 6 months
10. Hepatitis C+ or previous diagnosis of cirrhosis
11. Liver Function Studies great than or equal to triple of normal values

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological Male
Enrollment: 4 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2010-05-31 (Actual); Study Completion 2010-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Rollins, MD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No data are available for this study as the PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed.
Period: Overall Study
Arm/Group | Pioglitazone | Observation/Comparison
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No data are available for this study as the PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Observation/Comparison | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]
0 Participants

OUTCOME MEASURES:

1. Primary Outcome: Percent of Liver Fat Pre/Post Challenge With Daily Pioglitazone 45 mg
Description: No data are available for this study as the PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed
Time Frame: 16 weeks
Population: as for baseline characteristics
Arm/Group | Pioglitazone | Observation/Comparison
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Fine Needle Aspiration of Fat Pre/Post With Daily Pioglitazone 45 mg
Time Frame: 16 weeks
Population: Investigator left the university mid way through the study and unable to find him.
Arm/Group | Pioglitazone | Observation/Comparison
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No data are available for this study as the PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed
Description: No data are available for this study as the PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed
Arm/Group | Pioglitazone | Observation/Comparison
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes